CLINICAL TRIAL: NCT06866756
Title: Experience in Percutaneous Coronary Intervention With Sirolimus Drug-Coated Balloon and Paclitaxel Drug-Coated Balloon
Status: Recruiting | Type: Observational
Sponsor: Andres Iñiguez Romo (Other)
Responsible Party: Sponsor-Investigator, Andres Iñiguez Romo, Head of Cardiology Department, Fundacin Biomedica Galicia Sur
Organization: Fundacin Biomedica Galicia Sur (Other)
Other Study IDs: CAR-BAL-001
Record Dates: First submitted 2025-02-26; First posted 2025-03-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: DCB; Drug Coated Balloon; Drug eluting balloon; percutaneous coronary intervention; PCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sirolimus-Coated Balloon: Patients with coronary artery disease treated with Sirolimus-Coated Balloon
- Paclitaxel-Coated Balloon: Patients with coronary artery disease treated with Paclitaxel-Coated Balloon

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of mortality worldwide, with a significant burden in low- and middle-income countries. Acute coronary syndrome (ACS) is often the first clinical manifestation of CVD, representing a major cause of morbidity and mortality. Global variations exist in revascularization rates and long-term mortality following ACS. It is estimated that 12% of disability-adjusted life years are lost annually due to CVD. Drug-coated balloons (DCB) constitute a promising technology to overcome few disadvantages of current latest generation of drug-eluting stents (DES). The safety of these devices has been proven previously. However, there is few data regarding its efficacy in a broad spectrum of clinical setting and patient population.

Hypothesis:

The sirolimus-coated drug-eluting balloon demonstrates comparable safety and efficacy to the paclitaxel-coated balloon in patients undergoing angioplasty for coronary artery disease.

Primary Objective:

To assess the safety and efficacy of paclitaxel- vs. sirolimus-coated drug-eluting balloon over 12 months in patients undergoing coronary angioplasty for in-stent restenosis or small-vessel stenosis.

Secondary Objectives:

To compare the efficacy (freedom from target vessel failure) of both balloons at 12 months.

To evaluate the safety of paclitaxel- vs. sirolimus-coated balloon in coronary revascularization at 12 months.

Study Design:

Study Type: Prospective, single-center, analytical cohort study.

Population: Patients undergoing angioplasty with paclitaxel- or sirolimus-coated drug-eluting balloons according to standard clinical practice.

Inclusion Criteria: Patients with De novo lesion and in stent reestenosis.

Study Period: From September 2021 to September 2026 or until the required sample size is achieved.

Study Importance:

This study will provide comparative evidence on the use of paclitaxel- and sirolimus-coated DCBs in coronary revascularization. The findings may contribute to future clinical recommendations for the optimal use of DCBs in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with De novo lesion and in stent reestenosis.

Exclusion Criteria:

* The patient is not a candidate for balloon treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with coronary artery disease eligible for percutaneous coronary intervention with a balloon
Sampling Method: Probability Sample
Enrollment: 479 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Target lesions revascularization | 5 years
  Rate of clinically driven target lesion revascularization (TLR) at 12 months, defined as any repeat percutaneous intervention or surgical bypass of the target lesion due to symptoms or objective evidence of ischemia

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 5 years
  Incidence of Major Adverse Cardiovascular Events (MACE) at 5 years, defined as a composite of cardiovascular death, non-fatal myocardial infarction, and clinically driven lesion revascularization. Each event will be independently adjudicated by a clinical events committee.

CONTACTS AND LOCATIONS:
Overall Officials: Victor A Jimenez Diaz, MD, MPH, Principal Investigator — Servicio Galego de Saude. Hospital Álvaro Cunqueiro; Andres Iñiguez Romo, MD, PhD, Study Chair — Servicio Galego de Saude. Hospital Álvaro Cunqueiro
Locations (1):
- Hospital Álvaro Cunqueiro, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data used to support the findings of this study are available from the corresponding author upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Deidentified individual participant data and supporting documents will be available beginning 6 months after publication of the primary results and for a period of 5 years. Availability beyond this period will be considered upon request.
Access Criteria: Qualified researchers may request access to the deidentified IPD and supporting information for scientifically sound proposals. Access will be granted after approval by the principal investigator and the signing of a data use agreement. Data will be shared via secure transfer.